CLINICAL TRIAL: NCT03721445
Title: If Heart Rate Variability Can Predict Continuous Positive Airway Pressure Acceptance and Compliance for Patients With Obstructive Sleep Apnea ?
Brief Title: Could HRV be a Valuable Predictor for CPAP Adherence?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Mei-Chen Yang, Attending physician, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Other Study IDs: 07-XD-093
Record Dates: First submitted 2018-10-15; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: OSA; Autonomic Dysfunction; PAP; Adherence, Patient
MeSH Terms: conditions — Primary Dysautonomias; Patient Compliance | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CPAP opponent: CPAP opponent: moderate to severe OSA patients who refused CPAP therapy after PSG study and CPAP titration test.
- CPAP acceptor: CPAP acceptor: moderate to severe OSA patients who accepted CPAP therapy after PSG study and CPAP titration test and had purchased a PAP at home for long term use.
  Interventions: Device: continuous positive airway pressure

INTERVENTIONS:
Device: continuous positive airway pressure — Could the changes of HRV between PSG night and CPAP titration night predict the CPAP adherence?
  Groups: CPAP acceptor

SUMMARY:
This study aim to evaluate if the improvement of heart rate variability for the continuous positive airway pressure titration night can predict the short and long term continuous positive airway pressure adherence for patients with moderate to severe OSA.

DETAILED DESCRIPTION:
Heart rate variability (HRV) represents autonomic regulation and had been used in varies situation, especially the associated with cardiovascular outcomes and psychological diseases. HRV was also well known associated with the severity of obstructive sleep apnea (OSA) and could be improved after adequate treatments for OSA. Continuous positive airway pressure (CPAP) is the first choice of treatment for OSA and had been proved to able to improve HRV in OSA patients. However, the CPAP adherence is always problematic. Many CPAP predictors had been well documented but the HRV is never evaluated to be a potential predictor of CPAP adherence.

Therefore, this study will evaluate the changes of HRV for polysomnography (PSG) night, for CPAP titration night to see if the changes of HRV in the CPAP titration night could predict CPAP adherence for OSA patients in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. aged:20~75y/o
2. PSG revealed moderate to severe OSA (apnea hypopnea index [AHI] ≧15/hour)
3. had been completed CPAP titration test

Exclusion Criteria:

1. aged<20y/o or >75 y/o
2. mild OSA, (AHI <15/hour), or no OSA (AHI<5/hour)
3. unstable cardiopulmonary disease, psychological diseases, using sleep pills.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: moderate to severe OSA patients proved by PSG study and had been received CPAP titration test and had been prescribed CPAP therapy at home.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
If changes in LF/HF ratio (Low frequency/High frequency ratio) could be a valuable predictor for CPAP acceptance in OSA patients? | 1 month
  Changes of LF/HF ratio between PSG study night and CPAP titration night will be measured and evaluated its association with CPAP acceptance of one month CPAP trial at home in moderate to severe OSA patients.

SECONDARY OUTCOMES:
If CPAP treatment could improve LF/HF ratio after 6 months of treatment in moderate to severe OSA patients? | 6 months
  After CPAP treatments 6 months, PSG examination will be followed-up again. The changes of LF/HF ratio between baseline PSG and 6-months PSG will be measured and be evaluated it's differences between different CPAP usage pattern (no any use in CPAP opponents, suboptimal use in CPAP acceptors and optimal use in CPAP acceptors ).

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chen Yang, MD, Principal Investigator — Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (2):
- Taiwan (2):
  - Mei-Chen Yang, New Taipei City
  - Taipei Tzu-Chi Hospital, Buddhist Tzu-Chi Medical Foundation, New Taipei City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Noda A, Yasuma F, Okada T, Yokota M. Circadian rhythm of autonomic activity in patients with obstructive sleep apnea syndrome. Clin Cardiol. 1998 Apr;21(4):271-6. doi: 10.1002/clc.4960210408. PMID 9562937
- [Background] Palma JA, Iriarte J, Fernandez S, Alegre M, Valencia M, Artieda J, Urrestarazu E. Long-term continuous positive airway pressure therapy improves cardiac autonomic tone during sleep in patients with obstructive sleep apnea. Clin Auton Res. 2015 Aug;25(4):225-32. doi: 10.1007/s10286-015-0297-7. Epub 2015 May 23. PMID 26001693
- [Background] Walter LM, Biggs SN, Nisbet LC, Weichard AJ, Hollis SL, Davey MJ, Anderson V, Nixon GM, Horne RS. Improved long-term autonomic function following resolution of sleep-disordered breathing in preschool-aged children. Sleep Breath. 2016 Mar;20(1):309-19. doi: 10.1007/s11325-015-1268-x. Epub 2015 Oct 2. PMID 26432070
- [Background] Gong X, Huang L, Liu X, Li C, Mao X, Liu W, Huang X, Chu H, Wang Y, Wu W, Lu J. Correlation Analysis between Polysomnography Diagnostic Indices and Heart Rate Variability Parameters among Patients with Obstructive Sleep Apnea Hypopnea Syndrome. PLoS One. 2016 Jun 2;11(6):e0156628. doi: 10.1371/journal.pone.0156628. eCollection 2016. PMID 27253187
- [Background] Terziyski KV, Draganova AI, Taralov ZZ, Ilchev IS, Kostianev SS. The effect of continuous positive airway pressure on heart rate variability during the night in patients with chronic heart failure and central sleep apnoea. Clin Exp Pharmacol Physiol. 2016 Dec;43(12):1185-1190. doi: 10.1111/1440-1681.12662. PMID 27560005